CLINICAL TRIAL: NCT07042321
Title: Triglyceride Glucol Index for Predicting the Value of No-Reflow in Patients Undergoing Emergency PCI for Acute Myocardial Infarction
Brief Title: Risk Factors for Microvascular Obstruction Post-Emergency PCI in AMI Patients
Status: Recruiting | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yu Cao, Cardiology Professor, The Third Xiangya Hospital of Central South University
Other Study IDs: cy25231
Record Dates: First submitted 2025-05-28; First posted 2025-06-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Acute Myocardial Infarction (AMI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High TYG Index Group
- Medium TYG Index Group
- Low TYG Index Group

SUMMARY:
The goal of this prospective cohort study is to investigate the relationship between the TyG index and early identification of MVO in AMI patients undergoing emergency PCI and CMR imaging. The study will enroll approximately 300 AMI patients treated at Xiangya Third Hospital of Central South University from June 2024 to August 2025. The main questions it aims to answer are:

* How does the TyG index correlate with the early detection of MVO?
* What differences in cardiovascular adverse events during hospitalization exist between groups with varying TyG index levels? Participants will undergo emergency PCI and CMR imaging within 3-7 days post-procedure. Data collected will include demographic characteristics, clinical history, coronary angiography data, laboratory test indicators (especially metabolic markers such as blood glucose and lipids), IVUS-related plaque information, and CMR results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* STEMI symptom onset time < 12 hours.
* STEMI symptom onset time 12-48 hours, with ongoing ischemic symptoms, hemodynamic instability, or life-threatening ventricular arrhythmias.
* Very high-risk NSTEMI; undergoing emergency PCI treatment.
* Voluntary signed informed consent form.

Exclusion Criteria:

* Non-obstructive acute myocardial infarction.
* Severe chronic kidney disease (defined as estimated glomerular filtration rate <20 mL/min per 1.73 m²).
* Pregnant women or those planning to become pregnant.
* Failure of emergency PCI.
* Unclear CMR images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The presence or absence of microvascular obstruction (MVO) diagnosed by cardiac magnetic resonance (CMR) within 3-7 days postoperatively | 3-7 days postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Third Hospital of Central South University, Changsha, Hunan Province,China, China

IPD SHARING:
Plan to Share IPD: No
The nature of the data collected in this study includes sensitive information that is closely tied to the identity of the participants. Out of respect for the privacy and confidentiality of our participants, and in strict adherence to the terms of the informed consent they provided, we are unable to share individual participant data. We believe that protecting the privacy of our participants is of utmost importance, and we are committed to upholding these ethical standards throughout our research.

REFERENCES:
- [Result] Kim MK, Ahn CW, Kang S, Nam JS, Kim KR, Park JS. Relationship between the triglyceride glucose index and coronary artery calcification in Korean adults. Cardiovasc Diabetol. 2017 Aug 23;16(1):108. doi: 10.1186/s12933-017-0589-4. PMID 28830471
- [Result] Soeda T, Higuma T, Abe N, Yamada M, Yokoyama H, Shibutani S, Ong DS, Vergallo R, Minami Y, Lee H, Okumura K, Jang IK. Morphological predictors for no reflow phenomenon after primary percutaneous coronary intervention in patients with ST-segment elevation myocardial infarction caused by plaque rupture. Eur Heart J Cardiovasc Imaging. 2017 Jan;18(1):103-110. doi: 10.1093/ehjci/jev341. Epub 2016 Jan 22. PMID 26800769
- [Result] Alberti KG, Zimmet P, Shaw J; IDF Epidemiology Task Force Consensus Group. The metabolic syndrome--a new worldwide definition. Lancet. 2005 Sep 24-30;366(9491):1059-62. doi: 10.1016/S0140-6736(05)67402-8. No abstract available. PMID 16182882

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-02-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT07042321/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent Form (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT07042321/ICF_001.pdf
  • Informed Consent Form: Ethical approval document (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT07042321/ICF_002.pdf